CLINICAL TRIAL: NCT00715949
Title: Neurocognitive Evaluation of Minor Traumatic Brain Injury in the Hospitalized Pediatric Population
Brief Title: Neurocognitive Evaluation of Mild Traumatic Brain Injury in the Hospitalized Pediatric Population
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pittsburgh (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-11-4572
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Mild Traumatic Brain Injury; Concussion
Keywords: traumatic brain injury; pediatric; neurocognitive; concussion
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mild Traumatic Brain Injury (MTBI) admits: admitted pediatric patients with mild traumatic brain injury (concussion)
  Interventions: Other: Immediate Post-concussion Assessment and Cognitive Testing

INTERVENTIONS:
Other: Immediate Post-concussion Assessment and Cognitive Testing — ImPACT© utilizes a battery of neurocognitive tests to assess neurologic deficits.

SUMMARY:
Brain injuries from trauma are common in children, often resulting in death and disability. Most brain injuries are minor, yet their treatment can be challenging. Because there are many different scales used to characterize the severity of brain injury, there is no consensus regarding how to manage patients with minor brain injuries. Specifically, there is no agreement on recommendations regarding the safety of return to activities following injury. In young athletes with minor brain injuries (i.e. concussions) there is strong data suggesting that return to baseline neurologic function is often delayed by days or weeks. Children allowed to return to activities too soon may be at a higher risk for a second concussion, may delay recovery or, in rare cases, die. Researchers have designed a computer-based testing system (ImPACT©) to objectively test for neurologic deficits following injury. This test has been used primarily in athletes following a concussion but is also applicable to children with brain injuries from non-sports related traumas. We propose to utilize this testing in pediatric patients admitted to the hospital with minor brain injury. The test would be administered at the time of the hospitalization as well as in the outpatient trauma clinic at the time of routine follow up. The test would allow us to determine if there are neurologic deficits, potentially subclinical, in these brain injured patients and how quickly they recover from their injuries. If successful, the testing will likely be useful in other clinical settings such as the primary care office (e.g. pediatrician), specialty care office (e.g. sports medicine), or emergency room to determine if an injured child requires additional intervention.

DETAILED DESCRIPTION:
BACKGROUND

Head injuries are a frequent source of morbidity and the most common source of mortality in the pediatric trauma population. [1] It is estimated that head injuries result in more than 500,000 emergency department visits, 95,000 hospital admissions and 7,000 deaths in the pediatric age-groups. [1] Despite the magnitude of these numbers, they likely underestimate the problem, as many injured children are not brought to medical attention. Fortunately, most head injuries (75%) are classified as minor. [2] While major head injuries obviously pose a greater threat to life for the individual, the sheer volume of minor head injuries, as well as the potential for enduring neurologic sequelae, makes them a significant public health problem. Management of this large group of patients can be most challenging due to a lack of consensus in the health care community regarding the definition of minor traumatic brain injury, the ideal assessment modality for the injured child and recommendations for return to activity following a brain injury. Return to play recommendations have traditionally been based on the grade of concussion and the clinical exam. However given the large number of concussion grading scales in existence and the subtle nature of many of the neurologic deficits, standard recommendations have been lacking. Further still, the tremendous variability in time to full recovery exhibited by brain-injured children make generic guidelines naïve.

While the recovery from head injury in children is variable and difficult to predict, the desire to return to activity however, is near constant. Determining when it is safe to return to play is thus important. Recent literature has highlighted the perils of premature return to activities (most notably contact sports) for children with traumatic brain injury. [3-6] Dangers include prolongation of post-concussive symptoms, increased risk of recurrence of injury and death.[3-6] Further, these dangers may be more common in the younger athletes.[7] However, there is evidence that even non-contact, exertional activities may be detrimental if initiated too quickly. It was the observation of the First International Conference on Concussion in Sport that no previously published guidelines for management of concussion was adequate for assessment of all concussions. Further, they recognized the utility of neuropsychological testing in understanding the injury and determining management for the concussed patient. [8] Unfortunately, the majority of treating clinicians have few tools available to help determine when it is appropriate for the individual to return to activities. One such tool that has been used extensively and effectively in the head injured athlete is the Immediate Post concussion Assessment and Cognitive Testing (ImPACT©) program. This is an interactive software program originally designed to assess subjective and objective cognitive abilities of the head injured athlete. The program has been validated for use in sports-related concussion. [9, 10] Studies of concussed athletes have demonstrated a much slower return to baseline than previously had been appreciated. [11] Further, the younger athletes (high school vs. college or professional) were the slowest to return to the baseline. [7] This program has proven quite useful in determining the optimal time to return to activities in the population of head injured athletes by providing objective data upon which to base recommendations.

The same decisions facing clinicians treating children with sports related head injuries also exist for other non-sports related mechanisms (e.g. motor vehicle collisions, falls). Motor vehicle related causes and falls are the most common sources of traumatic brain injury in children. [12] Sports and recreation account for less than 10% of hospitalized minor traumatic brain injuries. Non-sports related traumatic brain injuries are often more severe but can be equally as difficult to assess. Anecdotal evidence collected by the researchers with the ImPACT© team suggests that the neurocognitive testing would be similarly efficacious in the assessment of non-sports related brain injured patients.

Utilizing a treatment algorithm that involves neurocognitive testing at the level of the individual is most likely to effectively determine the suitability to return to activities and the need for specialty intervention.

SPECIFIC AIMS

1. To assess the feasibility of inpatient bedside neurocognitive testing of pediatric patients with minor traumatic brain injury.
2. To establish if neurocognitive deficits exist, and to what extent, in the cohort of hospitalized pediatric patients with minor traumatic brain injury.
3. To document the timing and extent of recovery for pediatric traumatic brain injury through follow-up neurocognitive testing.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric blunt trauma patients (age 11-19 years) admitted for treatment of minor traumatic brain injury will be eligible for inclusion in the study. For the purposes of this study, mild traumatic brain injury will include patients with a Glasgow Coma Scale (GCS) of 14-15 upon arrival in the trauma receiving area. This may include those patients with and without abnormalities on head CT scans.
* Children will be included regardless of race, gender or ethnicity. The distribution of gender, race, and ethnicity is expected to reflect that of the trauma population at The Children's Hospital of Philadelphia

Exclusion Criteria:

* Patients with penetrating injuries as well as patients treated and released from the emergency room will be excluded.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric blunt trauma patients (age 11-19 years) admitted to The Children's Hospital of Philadelphia for treatment of mild traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Nance, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Nance ML, Polk-Williams A, Collins MW, Wiebe DJ. Neurocognitive evaluation of mild traumatic brain injury in the hospitalized pediatric population. Ann Surg. 2009 May;249(5):859-63. doi: 10.1097/SLA.0b013e3181a41ae5. PMID 19387313

RESULTS

PARTICIPANT FLOW:
Groups:
- Admitted Pediatric With MTBI: admitted pediatric patients with minor traumatic brain injury participating in computerized neurocognitive testing
Period: Overall Study
Arm/Group | Admitted Pediatric With MTBI
Started | 120 (4 dropped because could not finish first test)
Completed | 116 (116 patients completed first test)
Not Completed | 4
Not completed — could not finish first test | 4

BASELINE CHARACTERISTICS:
Groups:
- Admitted Pediatric With MTBI: admitted pediatric patients with minor traumatic brain injury
Arm/Group | Admitted Pediatric With MTBI
Number analyzed (Participants) | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 116
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 81
Region of Enrollment [Number; unit: participants]
  United States | 116

OUTCOME MEASURES:

1. Primary Outcome: The Feasibility of Inpatient Bedside Neurocognitive Testing of Pediatric Patients With Minor Traumatic Brain Injury.
Description: In this study, we demonstrated the feasibility of administering a previously validated, computer-based neurocognitive test battery in the inpatient setting. Participation numbers were determined by the ability of the participant to attend to and complete computerized neurocognitive testing while hospitalized with minor traumatic brain injury (MTBI).
Time Frame: Initial testing within 72 hours of injury and subsequent testing at approximately 2-3 weeks after injury. Subjects were offered the opportunity to also undergo testing at 3 months post-injury.
Population: Analysis population includes only subjects who completed computerized neurocognitive tests. 120 subjects began the study, however 4 dropped out because they were unable to complete the first test and were not included in the final number of analyzed participants.
Measure: Number; unit: participants
Arm/Group | Admitted Pediatric With MTBI
Number analyzed (Participants) | 120
participants | 120

2. Secondary Outcome: To Establish if Neurocognitive Deficits Exist, and to What Extent, in the Cohort of Hospitalized Pediatric Patients With Minor Traumatic Brain Injury.
Time Frame: study completion
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Admitted Pediatric With MTBI
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No